CLINICAL TRIAL: NCT04400526
Title: Development of a Community-based Network to Identify and Refer Drug Abusers in Hong Kong
Brief Title: Development of a Community-based Network for Drug Abusers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BDF 190003
Record Dates: First submitted 2020-05-13; First posted 2020-05-22 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2020-05

CONDITIONS: Adolescent
Keywords: Hidden drug abuse; Community-based network; Ambassadors; Brief intervention; Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: A video competition for anti-drug abuse (Other): Phase 1 aims to increase the public awareness of hazardous effects of drug abuses and existing resources available for drug abusers through a video competition. We will co-organize a video competition for anti-drug abuse with C.H.O.I.C.E. The competition will appeal to the participation of all children (aged 13-18) living in the four targeted districts.
  Interventions: Behavioral: A video competition
- Phase 2: Developing a community-based network (Other): Phase 2 aims to develop a community-based network through training anti-drug ambassadors (ADAs). We target to recruit a total of 150 children aged 13 - 18 as ADAs through secondary schools and community centres in the four targeted districts by sending invitation letters. The content of the workshop will be designed by our expert panel. The content of the workshop will include (1) hazardous effects of drug abuse especially less psychotropic drugs such as Cannabis, (2) signs and symptoms of drug abuse particularly less psychotropic drugs like Cannabis, (3) alternatives to drug abuse, (4) community resources available, and (5) how to refer drug abusers. Besides, all children will be taught to use the AWARD model for referrals in the workshop.
  Interventions: Behavioral: A training workshop
- Phase 3: A mass promotional campaign (Other): Phase 3 aims to engage the public to join the community-based network through anti-drug activities organized by anti-drug ambassadors. They are encouraged to design their own promotional activities for community members in the targeted districts.Types of activities can include but not limited to health talks, booths, outreaching activities, games, posters, leaflets and websites.
  Interventions: Behavioral: A mass promotional campaign

INTERVENTIONS:
Behavioral: A video competition — Each Individual/group will be required to produce a maximum of 2-minute video on one of the following themes: (1) the hazardous effects of drug especially less psychotropic drugs such as Cannabis, (2) encouraging messages to drug abusers, and (3) existing anti-drug services.
  Arms: Phase 1: A video competition for anti-drug abuse
Behavioral: A training workshop — The workshop will last for 6 hours, and will be delivered by an experienced counsellor from C.H.O.I.C.E. The content of the workshop will include (1) hazardous effects of drug abuse especially less psychotropic drugs such as Cannabis, (2) signs and symptoms of drug abuse particularly less psychotropic drugs like Cannabis, (3) alternatives to drug abuse, (4) community resources available, and (5) how to refer drug abusers. Besides, all children will be taught to use the AWARD model for referrals in the workshop.
  Arms: Phase 2: Developing a community-based network
Behavioral: A mass promotional campaign — Children who complete the training workshop in phase 2 will be invited to join phase 3. They are encouraged to design their own promotional activities for community members in the targeted districts. The activities can be delivered by a group (a maximum of 5 ADAs per group) or by an individual. Types of activities can include but not limited to health talks, booths, outreaching activities, games, posters, leaflets and websites. Likewise, if the ADAs encounter any drug abuser in their social circles, the ADAs will be asked to deliver a brief advice based on the AWARD model.
  Arms: Phase 3: A mass promotional campaign

SUMMARY:
Hidden drug abuse remains a significant concern for public health. An appropriate intervention is necessary to encourage hidden drug abusers to report their situations and seek professional help. This project aims to develop a community-based network to identify and refer hidden drug abusers in Hong Kong, and assess its effectiveness.

DETAILED DESCRIPTION:
This study will be completed within 18 months, and be divided into 3 Phases, including (1) a video competition for anti-drug abuse, (2) development of a community-based network through training 150 peers aged 13-18 as anti-drug ambassadors (ADAs) to deliver anti-drug messages based on the AWARD model, and (3) a mass promotional campaign organized by ADAs in the community. A one-group pre-test and repeated post-test design will be adopted to evaluate the overall effectiveness of the community-based network. We will assess the knowledge, attitudes and practices regarding anti-drug abuse of the ADAs. Data collection will be conducted at baseline, post-training, 3 months and 6 months after the training workshop.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 - 18 years
* Able to speak Cantonese and read Chinese

Exclusion Criteria:

* identified cognitive, behavioral or learning problem(s)
* identified mental illness(es)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge about the hazardous effects of drug abuse among ADAs by using Beat Drugs Fund Evaluation Question Set No. 2 | Immediately after the training workshop
  Change in knowledge about the hazardous effects of drug abuse among ADAs immediately after the training workshop when compared to baseline

SECONDARY OUTCOMES:
Change in knowledge about the hazardous effects of drug abuse among ADAs by using Beat Drugs Fund Evaluation Question Set No. 2 | 3 months after the training workshop
  Change in knowledge about the hazardous effects of drug abuse among ADAs at 3 months after the training workshop when compared to baseline
Change in knowledge about the hazardous effects of drug abuse among ADAs by using Beat Drugs Fund Evaluation Question Set No. 2 | 6 months after the training workshop
  Change in knowledge about the hazardous effects of drug abuse among ADAs at 6 months after the training workshop when compared to baseline
Change in attitudes towards drug abuse and anti-drug abuse among ADAs by using Beat Drugs Fund Evaluation Question Set No. 1 | Immediately after the training workshop
  Change in attitudes towards drug abuse and anti-drug abuse among ADAs immediately after the training workshop when compared to baseline
Change in attitudes towards drug abuse and anti-drug abuse among ADAs by using Beat Drugs Fund Evaluation Question Set No. 1 | 3 months after the training workshop
  Change in attitudes towards drug abuse and anti-drug abuse among ADAs at 3 months after the training workshop when compared to baseline
Change in attitudes towards drug abuse and anti-drug abuse among ADAs by using Beat Drugs Fund Evaluation Question Set No. 1 | 6 months after the training workshop
  Change in attitudes towards drug abuse and anti-drug abuse among ADAs at 6 months after the training workshop when compared to baseline
Change in anti-drug practices among ADAs by using Anti-Drug Practice Questionnaires | 3 months after the training workshop
  Personal development questions among ADAs at 3 months after the training workshop when compared to baseline
Change in anti-drug practices among ADAs by using Anti-Drug Practice Questionnaires | 6 months after the training workshop
  Personal development questions among ADAs at 6 months after the training workshop when compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Ka Yan HO, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No